CLINICAL TRIAL: NCT00275821
Title: A Randomized, Double-masked, Active-controlled, Multi-center Study Comparing the Efficacy and Safety of Ranibizumab Administered as Two Dosing Regimens in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Brief Title: Efficacy and Safety of Ranibizumab in Patients With Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration (AMD)
Acronym: EXCITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002A2302
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Results first posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-02

CONDITIONS: Age Related Macular Degeneration
Keywords: Age-related macular degeneration, ranibizumab
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Ranibizumab 0.3 mg - 3 times monthly, then quarterly (Experimental)
  Interventions: Drug: Ranibizumab 0.3 mg - 3 times monthly, then quarterly
- Ranibizumab 0.5 mg - 3 times monthly, then quarterly (Experimental)
  Interventions: Drug: Ranibizumab 0.5 mg - 3 times monthly, then quarterly
- Ranibizumab 0.3 mg monthly (Active Comparator)
  Interventions: Drug: Ranibizumab 0.3 mg monthly

INTERVENTIONS:
Drug: Ranibizumab 0.3 mg - 3 times monthly, then quarterly — Subjects received intravitreal injections (in the study eye) of ranibizumab 0.3 mg over a duration of 12 months. They were treated monthly for 3 consecutive months and then quarterly for the remainder of the study. On those months when ranibizumab was not administered, patients received a sham injection to preserve the masking of the treatment arms.
  Arms: Ranibizumab 0.3 mg - 3 times monthly, then quarterly
Drug: Ranibizumab 0.5 mg - 3 times monthly, then quarterly — Subjects received intravitreal injections (in the study eye) of ranibizumab 0.5 mg over a duration of 12 months. They were treated monthly for 3 consecutive months and then quarterly for the remainder of the study. On those months when ranibizumab was not administered, patients received a sham injection to preserve the masking of the treatment arms.
  Arms: Ranibizumab 0.5 mg - 3 times monthly, then quarterly
Drug: Ranibizumab 0.3 mg monthly — Subjects received monthly intravitreal injections (in the study eye) of ranibizumab 0.5 mg over a duration of 12 months. On those months when ranibizumab was not administered, patients received a sham injection to preserve the masking of the treatment arms.
  Arms: Ranibizumab 0.3 mg monthly

SUMMARY:
The study will test if the efficacy and safety of an alternative dosing regimen is as effective as monthly injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or recurrent subfoveal CNV secondary to AMD, including those with predominantly classic, minimally classic or occult lesions with no classic component
* Patients who have a BCVA score between 73 and 24 letters, inclusively, in the study eye using ETDRS-like grading charts (approximately 20/40 to 20/320)

Exclusion Criteria:

* Prior treatment in the study eye with verteporfin, external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, or transpupillary thermotherapy.
* History of submacular surgery or other surgical intervention for AMD in the study eye, glaucoma filtration surgery, corneal transplant surgery.
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within one month preceding Baseline.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2005-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis - Including Sites in Germany
Locations (1):
- Novartis, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab 0.3 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.5 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.3 mg Monthly
Started | 120 | 118 | 115
Completed | 106 | 95 | 103
Not Completed | 14 | 23 | 12
Not completed — Adverse Event | 4 | 12 | 5
Not completed — Administrative problems | 3 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Death | 0 | 2 | 1
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Protocol Violation | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.3 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.5 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.3 mg Monthly | Total
Number analyzed (Participants) | 120 | 118 | 115 | 353
Age, Customized [Number; unit: Participants]
  50 - < 65 | 13 | 12 | 10 | 35
  65 - < 75 | 37 | 28 | 45 | 110
  75 - < 85 | 61 | 72 | 46 | 179
  ≥ 85 | 9 | 6 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 73 | 66 | 209
  Male | 50 | 45 | 49 | 144

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best-corrected Visual Acuity of the Study Eye at Month 12
Description: Visual acuity (VA) was assessed in both eyes at each study visit using best correction determined from protocol refraction. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at an initial testing distance of 4 meters.
Time Frame: Baseline to Month 12
Population: Per-Protocol (PP) population includes a subset of patients from the Intent to Treat (ITT) population who completed Month 12/Visit 15, had an assessment of Best Corrected Visual Acuity in the study eye at Month 12/Visit 15 and did not have any major study protocol deviations.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab 0.3 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.5 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.3 mg Monthly
Number analyzed (Participants) | 104 | 88 | 101
letters | 4.9 (13.13) | 3.8 (13.33) | 8.3 (11.31)

2. Secondary Outcome: Mean Change From Baseline in the Total Lesion Area of the Study Eye at Month 12
Description: Fluorescein angiography was conducted in conjunction with color fundus photography at screening and at Months 6 and 12. Investigators used digital fluorescein angiograms to determine presence or absence of choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD).
Time Frame: Baseline to Month 12
Population: The intent to treat (ITT) population, with use of Last Observation Carried Forward (LOCF), consisted of all patients randomized into the study. Patients were analyzed according to the treatment group to which they were randomized. Only patients with available data at baseline and Month 12 were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Ranibizumab 0.3 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.5 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.3 mg Monthly
Number analyzed (Participants) | 113 | 105 | 108
mm^2 | -0.21 (5.616) | -1.51 (4.802) | -1.28 (4.367)

3. Secondary Outcome: Mean Change From Baseline in Retinal Thickness at the Central Point of the Study Eye at Month 12
Description: Optical Coherence Tomography (OCT) was performed on both eyes at screening and monthly from baseline through Month 12 prior to study drug administration. OCT images were evaluated at the central reading center (CRC) by trained graders and ophthalmologists experienced in clinical trials.
Time Frame: Baseline to Month 12
Population: Intent to Treat (ITT) population, with use of Last Observation Carried Forward (LOCF), consisted of all patients randomized into the study. Patients were analyzed according to the treatment group to which they were randomized. Only patients with available data at baseline and Month 12 were included in the analysis.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Ranibizumab 0.3 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.5 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.3 mg Monthly
Number analyzed (Participants) | 100 | 100 | 95
micrometers | -96.0 (96.82) | -105.6 (128.98) | -105.3 (128.55)

4. Secondary Outcome: Mean Change From Baseline in Retinal Thickness at the Central Subfield of the Study Eye at Month 12
Description: as for outcome 3
Time Frame: Baseline to Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micrometers
Arm/Group | Ranibizumab 0.3 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.5 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.3 mg Monthly
Number analyzed (Participants) | 100 | 100 | 95
Micrometers | -93.3 (100.88) | -97.5 (117.52) | -97.9 (112.47)

ADVERSE EVENTS:
Arm/Group | Ranibizumab 0.3 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.5 mg - 3 Times Monthly, Then Quarterly | Ranibizumab 0.3 mg Monthly
Serious Adverse Events (participants affected / at risk) | 15/120 | 23/118 | 20/115
Other Adverse Events (participants affected / at risk) | 66/120 | 71/118 | 64/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.3 mg - 3 Times Monthly, Then Quarterly (N=120) | Ranibizumab 0.5 mg - 3 Times Monthly, Then Quarterly (N=118) | Ranibizumab 0.3 mg Monthly (N=115)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2
Atrial flutter (Cardiac disorders) | 0 | 2 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Blindness transient (Study eye) (Eye disorders) | 0 | 1 | 0
Choroidal neovascularisation (Fellow eye) (Eye disorders) | 1 | 0 | 0
Retinal artery spasm (Study eye) (Eye disorders) | 1 | 0 | 0
Retinal detachment (Study eye) (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Study eye) (Eye disorders) | 0 | 1 | 0
Retinal pigment epithelial tear (Study eye) (Eye disorders) | 0 | 2 | 0
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Perianal abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1
Cataract traumatic (Study eye) (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Study eye) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Removal of internal fixation (Surgical and medical procedures) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.3 mg - 3 Times Monthly, Then Quarterly (N=120) | Ranibizumab 0.5 mg - 3 Times Monthly, Then Quarterly (N=118) | Ranibizumab 0.3 mg Monthly (N=115)
Blepharitis (Study eye) (Eye disorders) | 3 | 6 | 3
Choroidal neovascularisation (Fellow eye) (Eye disorders) | 7 | 6 | 3
Conjunctival haemorrhage (Study eye) (Eye disorders) | 23 | 19 | 12
Eye pain (Study eye) (Eye disorders) | 22 | 14 | 24
Eye pruritus (Study eye) (Eye disorders) | 1 | 3 | 6
Lacrimation increased (Study eye) (Eye disorders) | 4 | 1 | 6
Ocular hyperaemia (Study eye) (Eye disorders) | 8 | 10 | 7
Retinal haemorrhage (Study eye) (Eye disorders) | 4 | 8 | 2
Visual acuity reduced (Study eye) (Eye disorders) | 15 | 19 | 9
Vitreous floaters (Study eye) (Eye disorders) | 6 | 6 | 8
Nasopharyngitis (Infections and infestations) | 11 | 4 | 8
Intraocular pressure increased (Study eye) (Investigations) | 6 | 7 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 7
Headache (Nervous system disorders) | 2 | 6 | 5
Hypertension (Vascular disorders) | 10 | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.